CLINICAL TRIAL: NCT00276042
Title: Prospective, Randomized, Investigator-Blind Trial to Evaluate the Bacteriologic Eradication, Safety and Tolerability, and Pharmacokinetics of Different Dosages of Faropenem Medoxomil BID for 10 Days in the Treatment of Acute Otitis Media
Brief Title: A Trial to Evaluate Faropenem Medoxomil in the Treatment of Acute Otitis Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Replidyne (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REP-FAR-008
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Otitis Media
Keywords: AOM
MeSH Terms: conditions — Otitis Media | interventions — faropenem medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Faropenem Medoxomil

SUMMARY:
The study will be conducted in infants and children with acute otitis media, 6 months to less than 7 years old, in Costa Rica and Israel. The primary objective of this trial will be to describe bacteriologic efficacy in those with initial culture positive specimens with different dosages of faropenem

DETAILED DESCRIPTION:
The study will be conducted in infants and children with acute otitis media, 6 months to <7 years old, in Costa Rica and Israel. Faropenem is to be used as therapy for both simple and complicated AOM.

ELIGIBILITY:
Inclusion Criteria:

* Acute Otis Media

Exclusion Criteria:

* Any antibiotic for more than 24 hours (unless a treatment failure) within 7 days prior to enrollment

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate bacteriologic efficacy

SECONDARY OUTCOMES:
To describe investigator assessment of clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Roger M Echols, MD, Study Director — Replidyne, Inc.
Locations (2):
- Local Institution, San José, Costa Rica
- Local Institution, Beersheba, Israel